CLINICAL TRIAL: NCT02257125
Title: ArmeoSenso - Rewarding vs. Non-rewarding Therapy of Patients With Arm Impairments Based on Wearable Movement Sensors
Brief Title: ArmeoSenso - Reward
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Stopped due to futility considerations:
  Sample size calculations have assumed smaller effect sizes than considered relevant now.
Sponsor: Cereneo AG (Industry)
Collaborators: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EKNZ (LU) 13079
Record Dates: First submitted 2014-09-30; First posted 2014-10-06 (Estimated); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Stroke
Keywords: rehabilitation; virtual reality; stroke; upper extremity; arm; feedback; reward
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- high incentive (Experimental): game version including visual effects and monetary rewards
  Interventions: Behavioral: high incentive
- low incentive (Active Comparator): game version without visual effects or monetary rewards
  Interventions: Behavioral: low incentive

INTERVENTIONS:
Behavioral: high incentive — Subjects are required to use their arms in order to control a virtual arm on a computer screen to prevent meteors from destroying a planet. The game includes visual effects and monetary rewards.
  Arms: high incentive
Behavioral: low incentive — Subjects are required to use their arms in order to control a virtual "hand" on a computer screen to prevent objects from reaching the bottom. The game does not include visual effects or monetary rewards.
  Arms: low incentive

SUMMARY:
This study investigates the use of motivating/rewarding features in a computer based arm rehabilitation program. Half of the subjects will take part, besides receiving standard therapy, in a computer based program delivering a game like scenario with visual effects and monetary rewards in case of successful level completion, while the other half will take part in a similar program without visual effects or the possibility to earn money.

DETAILED DESCRIPTION:
Rewards not only increase motivation to train, but have also been shown to influence motor skill learning via activation of dopaminergic brain structures. In goal oriented tasks, receiving information about goal achievement has a rewarding value, which is further increased if performance has monetary consequences. Computer games often strengthen this kind of information by presenting explosions and other salient stimuli when a goal is achieved (e.g. a target has been reached). The current study investigates the outcome of an arm rehabilitation program, based on such a computer game delivered in two versions. Stroke patients are asked to use their impaired arms to perform goal oriented movements. Movements are translated into movements of a virtual arm on a computer screen. Goals are "meteors", threatening to destroy a planet on which they fall, if not caught by the virtual arm. One version of the computer game delivers state of the art graphics including a number of visual effects and, if the planet was protected successfully, information about a monetary reward, whereas the other version of the program delivers schematic graphic objects only. Training time and intensity are kept constant and outcome measures, including standard clinical motor assessments, are compared between the groups.

ELIGIBILITY:
Inclusion Criteria:

* stroke survivor (max. 100 days post-stroke)
* upper extremity motor deficits
* patient can lift the paretic arm against gravity
* patient can move the hand at least 20x20 cm in a horizontal plane
* patient is able and willing to participate
* patient has signed informed consent

Exclusion Criteria:

* severe aphasia (impairing verbal instructions)
* severe dementia (impairing the capability to understand instructions)
* severe depression (impairing motivation to train)
* relevant (in the judgement of the investigator) impairment of visual perception, (impairing perception of goals and feedback on the computer screen)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-01-27 (Actual); Primary Completion 2019-10-28 (Actual); Study Completion 2019-10-28 (Actual)

PRIMARY OUTCOMES:
Change in ArmeoSenso - hand workspace | Assessed for each training visit (i.e., 15 visits over 3 weeks between day 2 and day 22): Main outcome is the change in hand workspace over the training intervention.
  The subject moves the affected arm as far as possible in all directions while sitting in a gaming position. Movement range is recorded.

SECONDARY OUTCOMES:
Motivation questionnaire | Assessed for each training visit (i.e., 15 visits over 3 weeks between day 2 and day 22)
  Measures motivation to train.
Wolf Motor Function Test | Baseline (day 1), post-training (day 23 ± 5 days) and 3 months post-training (day 113 ± 7 days); training lasts for 3 weeks (15 visits, one per workday)
  Quantifies upper extremity motor ability through timed and functional tasks.
Fugl-Meyer Assessment Upper Extremity | Baseline (day 1), post-training (day 23 ± 5 days) and 3 months post-training (day 113 ± 7 days); training lasts for 3 weeks (15 visits, one per workday)
  Measures motor impairment.
Box and Blocks Test | Baseline (day 1), post-training (day 23 ± 5 days) and 3 months post-training (day 113 ± 7 days); training lasts for 3 weeks (15 visits, one per workday)
  Measures gross manual dexterity.
ArmeoSenso: pointing task | Assessed for each training visit (i.e., 15 visits over 3 weeks between day 2 and day 22)
  Goal is to reach targets in the transversal plane in front of the subject: number of targets and time.
Motor Activity Log 14 (MAL-14) | Baseline (day 1), post-training (day 23 ± 5 days) and 3 months post-training (day 113 ± 7 days); training lasts for 3 weeks (15 visits, one per workday)
  Self-reported movement ability.
Barthel Index | Baseline (day 1), post-training (day 23 ± 5 days) and 3 months post-training (day 113 ± 7 days); training lasts for 3 weeks (15 visits, one per workday)
  Measure of independence in daily living.
NIHSS | Baseline (day 1), post-training (day 23 ± 5 days) and 3 months post-training (day 113 ± 7 days); training lasts for 3 weeks (15 visits, one per workday)
  Measure of stroke severity.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Luft, Prof., Principal Investigator — University of Zurich, University Hospital Zurich
Locations (3):
- Switzerland (3):
  - Cereneo, Center For Rehabilitation and Neurology, Vitznau, Canton of Lucerne
  - Klinik Adelheid, Unterägeri, Canton of Zug
  - Zuercher Reha Zentrum Wald, Wald

REFERENCES:
- [Derived] Widmer M, Held JPO, Wittmann F, Valladares B, Lambercy O, Sturzenegger C, Palla A, Lutz K, Luft AR. Reward During Arm Training Improves Impairment and Activity After Stroke: A Randomized Controlled Trial. Neurorehabil Neural Repair. 2022 Feb;36(2):140-150. doi: 10.1177/15459683211062898. Epub 2021 Dec 22. PMID 34937456
- [Derived] Widmer M, Held JP, Wittmann F, Lambercy O, Lutz K, Luft AR. Does motivation matter in upper-limb rehabilitation after stroke? ArmeoSenso-Reward: study protocol for a randomized controlled trial. Trials. 2017 Dec 2;18(1):580. doi: 10.1186/s13063-017-2328-2. PMID 29197412